CLINICAL TRIAL: NCT01601184
Title: An International, Randomized, Open-label Phase I/II Study of Vismodegib in Combination With Temozolomide Versus Temozolomide Alone in Adult Patients With Recurrent or Refractory Medulloblastomas Presenting an Activation of the Sonic Hedgehog (SHH) Pathway
Brief Title: Study of Vismodegib in Combination With Temozolomide Versus Temozolomide Alone in Patients With Medulloblastomas With an Activation of the Sonic Hedgehog Pathway
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The number of successes is not reached at the end of first stage of the phase II. The study is stopped.
Sponsor: Centre Leon Berard (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEVITEM; 2011-003372-37 (EudraCT Number)
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Histologically Confirmed Medulloblastoma; Activation of the Sonic Hedgehog (SHH) Pathway
Keywords: medulloblastoma; sonic hedgehog pathway; vismodegib
MeSH Terms: conditions — Microphthalmia, Isolated, with Coloboma 5; Medulloblastoma | interventions — HhAntag691; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- combination of vismodegib with temozolomide (Experimental): In the first step of the study (Phase I), 9 adult patients with relapsing or refractory medulloblastoma will be randomized (randomization ratio 2:1) to receive
  - Arm A: the combination of vismodegib (150 mg/day continuously) with temozolomide (150 mg/m2 during Cycle 1 [day 1 to day 5/ 28 day-cycle] and 200 mg/m2 during subsequent cycles) (6 patients)
  Interventions: Drug: vismodegib; Drug: Temozolomide
- temozolomide alone (Active Comparator): In the first step of the study (Phase I), 9 adult patients with relapsing or refractory medulloblastoma will be randomized (randomization ratio 2:1) to receive Arm B: temozolomide alone (150 mg/m2 day1 to day 5/ 28 day-cycle during Cycle 1 and 200 mg/m2 day 1 to day 5/ 28 day-cycle during subsequent cycles) (3 patients).
  Interventions: Drug: Temozolomide
- vismodegib alone (Other): Considering the rarity of the disease, the few therapeutic options available and the promising results reported with vismodegib in adult medulloblastoma : the Sponsor will consider (on case by case basis) the enrolment of patients previously treated by temozolomide in a 3rd independent and parallel study arm
  Interventions: Drug: vismodegib

INTERVENTIONS:
Drug: vismodegib — Hedgehog pathway antagonist Dosage: 150 mg orally with or without food at the same time every day
  Arms: combination of vismodegib with temozolomide; vismodegib alone
Drug: Temozolomide — alkylating agent Dosage: Dose in Cycle 1 is 150 mg/m2 orally once daily for 5 days followed by 23 days without treatment. At the start of Cycle 2, the dose is escalated to 200mg/m2 orally once daily for 5 days
  Other Names: temodal
  Arms: combination of vismodegib with temozolomide; temozolomide alone

SUMMARY:
The purpose of this study is to evaluate the safety of vismodegib in combination with temozolomide (primary objective - phase I) and to estimate the efficacy of vismodegib in combination with temozolomide in adult patients with recurrent, progressive, or refractory medulloblastomas to standard therapy measured by the 6-month progression-free rate (phase II).

This study is an open-label Phase I/II, international, randomized.

38 patients will be included in the study.

DETAILED DESCRIPTION:
Secondary objectives are :

phase I : to collect preliminary results on the 6-month progression-free rate of the combination vismodegib + temozolomide

PHASE II

To estimate in the two study arms:

* the objective response rate (Complete response + Partial Response according to WHO criteria) after 6 months of treatment
* the duration of treatment response
* the best overall response obtained during the study
* the progression-free survival (PFS)
* the time to progression (TTP)
* the time to treatment failure (TTF)
* In the combination arm (vismodegib + temozolomide): to further evaluate the safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients must have histologically confirmed medulloblastoma (including posterior fossa primitive neuroectodermal tumor) for which no known curative therapy exists
* Patients must have recurrent or refractory disease
* Patients must have evidence of measurable disease or lesion in pre-inclusion MRI. Patients with measurable spinal disease are eligible. NB: Patients with complete resection for recurrence are not eligible.
* Activation of the SHH pathway validated by IHC.
* ECOG performance status 0, 1 or 2
* Life expectancy ≥ 12 weeks
* Patients must have normal organ and marrow function as defined below:

Neutrophils ≥ 1. 5 G/L Platelets ≥ 100 G /L Hemoglobin ≥ 10g/dL Creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula or MDRD formula for patients older than 65 years ) or serum creatinine within normal limits or less than 1.5 x upper limit of normal (ULN) Total bilirubin ≤ 1.5 ULN ALAT and ASAT ≤ 2.5 ULN Serum albumin ≥ 25 g/L.

* Patients recovered from prior treatment-related toxicity (persistent treatment related toxicity <Grade 2 are allowed (NCI-CTCAE v4.0).
* Prior therapy:

No prior hedgehog antagonist vismodegib or other antagonists of the hedgehog pathway, and no prior temozolomide treatment for patients to be randomized in Arm A or B. Patients previously treated with temozolomide are eligible for enrollment in study arm C on a case by case basis and following sponsor agreement More than 4 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosoureas, 6 months after high dose therapy) or immunotherapy At least 3 months since prior craniospinal irradiation (≥ 23 Gy) At least 8 weeks since prior local irradiation to primary tumor At least 2 weeks since prior focal irradiation for symptomatic metastatic sites.

At least 1 week since prior colony-stimulating factors (e.g., G-CSF, GM-CSF, or erythropoietin)

* Women of childbearing potential* are required to have a negative serum pregnancy test within 72 hours prior to study treatment initiation (i.e. Cycle 1 Day 1).

  *: Female patients who meet at least one of the following criteria are defined as women of non-childbearing potential:

  ≥50 years old and naturally amenorrheic for ≥ 1 year Permanent premature ovarian failure confirmed by a specialist gynaecologist Previous bilateral salpingo-oophorectomy XY genotype, Turner's syndrome, or uterine agenesis Female patient who do not meet at least of the above criteria are defined as women of childbearing potential.
* An embryo-fetal development study in rats has confirmed the teratogenic potential of vismodegib. Therefore, women of child-bearing potential and men must use two forms of effective contraception (including one barrier method- refer to Appendix 4 for acceptable method of contraception) at least 4 weeks prior to study entry, during the study period and for at least 24 months post-treatment for women and 2 months post-treatment for men. Prior to dispensing vismodegib, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of vismodegib.
* Ability to understand and willingness to comply to follow-up visits.
* Covered by a medical insurance (in countries where applicable)

Exclusion Criteria:

* Tumor tissue sample not available for biological studies (from the initial diagnosis and/or relapse)
* Pregnant or breastfeeding women are not eligible.
* History of allergic reactions attributed to compounds of similar chemical composition to vismodegib.
* Any contraindications to temozolomide treatment as per Temodal® SPC (see Appendix 5).
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption. Patients must be able to swallow capsules.
* Uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia, defined as less than the lower limit of normal despite adequate electrolyte supplementation.
* History of congestive heart failure.
* History of ventricular arrhythmia requiring medication.
* Congenital long QT syndrome.
* Clinically significant unrelated systemic illness (e.g., serious infection or significant cardiac, pulmonary, hepatic, or other organ dysfunction) that would compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results.
* Patients using prohibited concomitant and/or concurrent medications (see section "Prohibited concomitant/concurrent treatments.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-06; Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of a fixed dose of vismodegib in combination with (phase I)temozolomide in adult patients with recurrent, progressive, or refractory to standard therapy medulloblastoma | during the first three months follow up
  number of severe toxicities occurring during the first 3 months of follow-up :
  * Toxic death
  * Grade 4 toxicity
  * Any grade 3 AE leading to study treatment interruption for more than 7 days or discontinuation.
To estimate the efficacy of vismodegib in combination with temozolomide in adult patients with recurrent, progressive, or refractory to standard therapy medulloblastoma (phase II) | 6 months after start of treatment
  the 6-month progression-free rate

SECONDARY OUTCOMES:
To collect preliminary results on the 6-month progression-free rate of the combination vismodegib + temozolomide (phase I) | 6 months after start of treatment
  measurement of progression free rate
To estimate in the two study arms the objective response rate after 6 months of treatment (phase II) | after 6 months of treatment
  measure by objective response rate
To estimate in the two study arms the duration of treatment response (phase II) | one year
  treatment response
To estimate in the two study arms the best overall response obtained during the study (phase II) | one year
To estimate in the two study arms the progression-free survival (PFS)(phase II) | one year
  measure of progression free rate
To estimate in the two study arms the time to treatment failure (phase II) | one year
frequency of adverse events based on the common toxicity criteria (CTC-AE-V4.0) grade | one year
  In the combination arm (vismodegib + temozolomide): to further evaluate the safety of the combination

CONTACTS AND LOCATIONS:
Overall Officials: didier frappaz, Principal Investigator — Centre Léon Bérard, Lyon
Locations (15):
- France (10):
  - CHU La Timone, Marseille, Bouches Du Rhône
  - Institut Claudius Régaud (iuct-oncopole), Toulouse, Haute-Garonne
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain, Loire Atlantique
  - Hopital Central de Nancy, Nancy, Meurthe Et Moselle
  - CHBS Hôpital du Scorff, Lorient, Morbihan
  - CHRU de Lille, Lille, Nord
  - Centre Léon Bérard, Lyon, Rhone
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Hopital de La Pitié Salpétrière, Paris, Île-de-France Region
- Italy (2):
  - BELLARIA Ospedale, Bologna
  - University of Turin, Torino
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - University Hospital Zurich, Zurich
- University College London Hospital - Mount Vernon Cancer Centre - Mount Vernon hospital, London, United Kingdom

REFERENCES:
- [Background] Lupi O. Correlations between the Sonic Hedgehog pathway and basal cell carcinoma. Int J Dermatol. 2007 Nov;46(11):1113-7. doi: 10.1111/j.1365-4632.2007.03391.x. PMID 17988327
- [Background] Romer JT, Kimura H, Magdaleno S, Sasai K, Fuller C, Baines H, Connelly M, Stewart CF, Gould S, Rubin LL, Curran T. Suppression of the Shh pathway using a small molecule inhibitor eliminates medulloblastoma in Ptc1(+/-)p53(-/-) mice. Cancer Cell. 2004 Sep;6(3):229-40. doi: 10.1016/j.ccr.2004.08.019. PMID 15380514
- [Background] Yauch RL, Gould SE, Scales SJ, Tang T, Tian H, Ahn CP, Marshall D, Fu L, Januario T, Kallop D, Nannini-Pepe M, Kotkow K, Marsters JC, Rubin LL, de Sauvage FJ. A paracrine requirement for hedgehog signalling in cancer. Nature. 2008 Sep 18;455(7211):406-10. doi: 10.1038/nature07275. Epub 2008 Aug 27. PMID 18754008
- [Background] Cornu P, Chatellier G, Fauchon F, Foncin JF, Faillot T, Dorwling-Carter D, Philippon J. [The prognosis of medulloblastoma in adults]. Neurochirurgie. 1990;36(4):218-24. French. PMID 2277658
- [Background] Coulbois S, Civit T, Grignon Y, Taillandier L, Girard F, Marchal C, Pinelli C, Auque J. [Adult medulloblastoma. Review of 22 patients]. Neurochirurgie. 2001 Feb;47(1):6-12. French. PMID 11283450
- [Background] Giordana MT, Schiffer P, Lanotte M, Girardi P, Chio A. Epidemiology of adult medulloblastoma. Int J Cancer. 1999 Mar 1;80(5):689-92. doi: 10.1002/(sici)1097-0215(19990301)80:53.0.co;2-g. PMID 10048968
- [Background] Brandes AA, Palmisano V, Monfardini S. Medulloblastoma in adults: clinical characteristics and treatment. Cancer Treat Rev. 1999 Feb;25(1):3-12. doi: 10.1053/ctrv.1998.0096. PMID 10212586
- [Background] Chan AW, Tarbell NJ, Black PM, Louis DN, Frosch MP, Ancukiewicz M, Chapman P, Loeffler JS. Adult medulloblastoma: prognostic factors and patterns of relapse. Neurosurgery. 2000 Sep;47(3):623-31; discussion 631-2. doi: 10.1097/00006123-200009000-00018. PMID 10981749
- [Background] del Charco JO, Bolek TW, McCollough WM, Maria BL, Kedar A, Braylan RC, Mickle JP, Buatti JM, Mendenhall NP, Marcus RB Jr. Medulloblastoma: time-dose relationship based on a 30-year review. Int J Radiat Oncol Biol Phys. 1998 Aug 1;42(1):147-54. doi: 10.1016/s0360-3016(98)00197-7. PMID 9747832
- [Background] Duffner PK. Long-term effects of radiation therapy on cognitive and endocrine function in children with leukemia and brain tumors. Neurologist. 2004 Nov;10(6):293-310. doi: 10.1097/01.nrl.0000144287.35993.96. PMID 15518596
- [Background] Padovani L, Sunyach MP, Perol D, Mercier C, Alapetite C, Haie-Meder C, Hoffstetter S, Muracciole X, Kerr C, Wagner JP, Lagrange JL, Maire JP, Cowen D, Frappaz D, Carrie C. Common strategy for adult and pediatric medulloblastoma: a multicenter series of 253 adults. Int J Radiat Oncol Biol Phys. 2007 Jun 1;68(2):433-40. doi: 10.1016/j.ijrobp.2006.12.030. PMID 17498567
- [Background] Abacioglu U, Uzel O, Sengoz M, Turkan S, Ober A. Medulloblastoma in adults: treatment results and prognostic factors. Int J Radiat Oncol Biol Phys. 2002 Nov 1;54(3):855-60. doi: 10.1016/s0360-3016(02)02986-3. PMID 12377339
- [Background] Carrie C, Lasset C, Alapetite C, Haie-Meder C, Hoffstetter S, Demaille MC, Kerr C, Wagner JP, Lagrange JL, Maire JP, et al. Multivariate analysis of prognostic factors in adult patients with medulloblastoma. Retrospective study of 156 patients. Cancer. 1994 Oct 15;74(8):2352-60. doi: 10.1002/1097-0142(19941015)74:83.0.co;2-h. PMID 7922986
- [Background] Evans AE, Jenkin RD, Sposto R, Ortega JA, Wilson CB, Wara W, Ertel IJ, Kramer S, Chang CH, Leikin SL, et al. The treatment of medulloblastoma. Results of a prospective randomized trial of radiation therapy with and without CCNU, vincristine, and prednisone. J Neurosurg. 1990 Apr;72(4):572-82. doi: 10.3171/jns.1990.72.4.0572. PMID 2319316
- [Background] Packer RJ, Sutton LN, Elterman R, Lange B, Goldwein J, Nicholson HS, Mulne L, Boyett J, D'Angio G, Wechsler-Jentzsch K, et al. Outcome for children with medulloblastoma treated with radiation and cisplatin, CCNU, and vincristine chemotherapy. J Neurosurg. 1994 Nov;81(5):690-8. doi: 10.3171/jns.1994.81.5.0690. PMID 7931615
- [Background] Packer RJ, Gajjar A, Vezina G, Rorke-Adams L, Burger PC, Robertson PL, Bayer L, LaFond D, Donahue BR, Marymont MH, Muraszko K, Langston J, Sposto R. Phase III study of craniospinal radiation therapy followed by adjuvant chemotherapy for newly diagnosed average-risk medulloblastoma. J Clin Oncol. 2006 Sep 1;24(25):4202-8. doi: 10.1200/JCO.2006.06.4980. PMID 16943538
- [Background] Tait DM, Thornton-Jones H, Bloom HJ, Lemerle J, Morris-Jones P. Adjuvant chemotherapy for medulloblastoma: the first multi-centre control trial of the International Society of Paediatric Oncology (SIOP I). Eur J Cancer. 1990 Apr;26(4):464-9. PMID 2141512
- [Background] Zeltzer PM, Boyett JM, Finlay JL, Albright AL, Rorke LB, Milstein JM, Allen JC, Stevens KR, Stanley P, Li H, Wisoff JH, Geyer JR, McGuire-Cullen P, Stehbens JA, Shurin SB, Packer RJ. Metastasis stage, adjuvant treatment, and residual tumor are prognostic factors for medulloblastoma in children: conclusions from the Children's Cancer Group 921 randomized phase III study. J Clin Oncol. 1999 Mar;17(3):832-45. doi: 10.1200/JCO.1999.17.3.832. PMID 10071274
- [Background] Riffaud L, Saikali S, Leray E, Hamlat A, Haegelen C, Vauleon E, Lesimple T. Survival and prognostic factors in a series of adults with medulloblastomas. J Neurosurg. 2009 Sep;111(3):478-87. doi: 10.3171/2009.1.JNS081004. PMID 19231932
- [Background] Nicholson HS, Kretschmar CS, Krailo M, Bernstein M, Kadota R, Fort D, Friedman H, Harris MB, Tedeschi-Blok N, Mazewski C, Sato J, Reaman GH. Phase 2 study of temozolomide in children and adolescents with recurrent central nervous system tumors: a report from the Children's Oncology Group. Cancer. 2007 Oct 1;110(7):1542-50. doi: 10.1002/cncr.22961. PMID 17705175
- [Background] Barone G, Maurizi P, Tamburrini G, Riccardi R. Role of temozolomide in pediatric brain tumors. Childs Nerv Syst. 2006 Jul;22(7):652-61. doi: 10.1007/s00381-006-0081-z. Epub 2006 Mar 25. PMID 16565851
- [Background] Kenney AM, Rowitch DH. Sonic hedgehog promotes G(1) cyclin expression and sustained cell cycle progression in mammalian neuronal precursors. Mol Cell Biol. 2000 Dec;20(23):9055-67. doi: 10.1128/MCB.20.23.9055-9067.2000. PMID 11074003
- [Background] Ingham PW, McMahon AP. Hedgehog signaling in animal development: paradigms and principles. Genes Dev. 2001 Dec 1;15(23):3059-87. doi: 10.1101/gad.938601. No abstract available. PMID 11731473
- [Background] Hooper JE, Scott MP. Communicating with Hedgehogs. Nat Rev Mol Cell Biol. 2005 Apr;6(4):306-17. doi: 10.1038/nrm1622. PMID 15803137
- [Background] Ferretti E, De Smaele E, Di Marcotullio L, Screpanti I, Gulino A. Hedgehog checkpoints in medulloblastoma: the chromosome 17p deletion paradigm. Trends Mol Med. 2005 Dec;11(12):537-45. doi: 10.1016/j.molmed.2005.10.005. Epub 2005 Nov 14. PMID 16290230
- [Background] Scales SJ, de Sauvage FJ. Mechanisms of Hedgehog pathway activation in cancer and implications for therapy. Trends Pharmacol Sci. 2009 Jun;30(6):303-12. doi: 10.1016/j.tips.2009.03.007. Epub 2009 May 13. PMID 19443052
- [Background] Rubin LL, de Sauvage FJ. Targeting the Hedgehog pathway in cancer. Nat Rev Drug Discov. 2006 Dec;5(12):1026-33. doi: 10.1038/nrd2086. PMID 17139287
- [Background] Pasca di Magliano M, Hebrok M. Hedgehog signalling in cancer formation and maintenance. Nat Rev Cancer. 2003 Dec;3(12):903-11. doi: 10.1038/nrc1229. No abstract available. PMID 14737121
- [Background] Von Hoff DD, LoRusso PM, Rudin CM, Reddy JC, Yauch RL, Tibes R, Weiss GJ, Borad MJ, Hann CL, Brahmer JR, Mackey HM, Lum BL, Darbonne WC, Marsters JC Jr, de Sauvage FJ, Low JA. Inhibition of the hedgehog pathway in advanced basal-cell carcinoma. N Engl J Med. 2009 Sep 17;361(12):1164-72. doi: 10.1056/NEJMoa0905360. Epub 2009 Sep 2. PMID 19726763
- [Background] Rudin CM, Hann CL, Laterra J, Yauch RL, Callahan CA, Fu L, Holcomb T, Stinson J, Gould SE, Coleman B, LoRusso PM, Von Hoff DD, de Sauvage FJ, Low JA. Treatment of medulloblastoma with hedgehog pathway inhibitor GDC-0449. N Engl J Med. 2009 Sep 17;361(12):1173-8. doi: 10.1056/NEJMoa0902903. Epub 2009 Sep 2. PMID 19726761
- [Background] Ellison DW, Dalton J, Kocak M, Nicholson SL, Fraga C, Neale G, Kenney AM, Brat DJ, Perry A, Yong WH, Taylor RE, Bailey S, Clifford SC, Gilbertson RJ. Medulloblastoma: clinicopathological correlates of SHH, WNT, and non-SHH/WNT molecular subgroups. Acta Neuropathol. 2011 Mar;121(3):381-96. doi: 10.1007/s00401-011-0800-8. Epub 2011 Jan 26. PMID 21267586
- [Background] Schwalbe EC, Lindsey JC, Straughton D, Hogg TL, Cole M, Megahed H, Ryan SL, Lusher ME, Taylor MD, Gilbertson RJ, Ellison DW, Bailey S, Clifford SC. Rapid diagnosis of medulloblastoma molecular subgroups. Clin Cancer Res. 2011 Apr 1;17(7):1883-94. doi: 10.1158/1078-0432.CCR-10-2210. Epub 2011 Feb 16. PMID 21325292
- [Background] Steg A, Vickers SM, Eloubeidi M, Wang W, Eltoum IA, Grizzle WE, Saif MW, Lobuglio AF, Frost AR, Johnson MR. Hedgehog pathway expression in heterogeneous pancreatic adenocarcinoma: implications for the molecular analysis of clinically available biopsies. Diagn Mol Pathol. 2007 Dec;16(4):229-37. doi: 10.1097/PDM.0b013e31811edc7e. PMID 18043287